CLINICAL TRIAL: NCT04613986
Title: Randomized, Prospective, Open-label, Controlled Parallel-group Trial Investigating the Efficacy of Therapeutic Plasma Exchange as an Adjunctive Strategy to Treat the Systemic Inflammatory Response Against SARS-CoV2 and the Associated Coagulopathy
Brief Title: Therapeutic Plasma Exchange as an Adjunctive Strategy to Treat Coagulopathy and Inflammation in Severe Covid-19
Acronym: PExCoV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SD01
Record Dates: First submitted 2020-11-02; First posted 2020-11-03 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Severe Covid-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard (No Intervention): Standard of care according to our current in house SOP
- Treatment (Experimental): Standard of care according to our current in house SOP + Therapeutic Plasmaexchange (d1, 3, 5)
  Interventions: Device: therapeutic plasmaexchnage

INTERVENTIONS:
Device: therapeutic plasmaexchnage — established method to exchange plasma (in order to remove injurious disease mediators, e.g. antibodies) or to replace consumed factors (e.g. vWF cleaving proteases)
  Arms: Treatment

SUMMARY:
Randomized controlled trial to analyse adjuvant therapeutic plasma exchange (TPE) in severe Covid-19 associated coagulopathy and systemic inflammation compared to current standard of care (SOC).

A total of three TPEs (d1, 3, 5) will be performed in the intervention group. Primary endpoint is the reversibility of relative ADAMTS13 deficiency (indicated by the change in ADAMTS13 / VWF:Ag ratio from day 1 to 7).

ELIGIBILITY:
Inclusion Criteria:

* Proven SARS-CoV2 infection
* Severe Covid-19 (indicated by respiratory failure requiring invasive mechanical ventilation)
* Evidence of coagulopathy (indicated by D-dimer > 10 mg/L)
* Evidence of systemic inflammation (CRP > 100 mg/L , ferritin > 500 ng/mL)

Exclusion Criteria:

* • Participation in another study with investigational drug within the 30 days preceding and during the present study,

  * Previous enrolment into the current study.
  * Extra corporeal membrane oxygenation (ECMO)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
relative ADAMTS13 deficiency | day 1 to 7
  ADAMTS13 / VWF:Ag